CLINICAL TRIAL: NCT00553787
Title: A Phase III Randomized, Double-Blind, Placebo Controlled Multicenter Study to Determine the Safety and Efficacy of VI-0521 in the Treatment of Obesity in Adults With Obesity-Related Co-Morbid Conditions
Brief Title: Study of VI-0521 Compared to Placebo in Treatment of Diabetes and Obesity in Adults With Obesity-Related Co-Morbid Conditions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OB-303
Record Dates: First submitted 2007-11-03; First posted 2007-11-06 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity, Type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VI-0521 Top (Experimental): high dose experimental treatment
  Interventions: Drug: VI-0521
- VI-0521 Mid (Experimental): mid dose experimental treatment
  Interventions: Drug: VI-0521
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: VI-0521

INTERVENTIONS:
Drug: VI-0521 — phentermine 15 mg and topiramate 92 mg, po once daily
  Arms: VI-0521 Top
Drug: VI-0521 — phentermine 7.5 mg and topiramate 46 mg, po once daily
  Arms: VI-0521 Mid
Drug: VI-0521 — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VI0521 compared to placebo in treatment of obesity in an adult population with obesity related co-morbid conditions.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* BMI ≥ 27 (no lower BMI limit for Type 2 diabetics)
* 70 years of age or less
* Have 2 or more of the following obesity-related co-morbid conditions:

  * Systolic blood pressure 140-160 mmHg (130-160 if diabetic);
  * Diastolic blood pressure 90-100 mmHg (85-100 if diabetic);
  * Requirement for 2 or more medications to achieve control (<140/90 mmHg)
* Triglyceride level between 200-400 mg/dL or requirement for 2 or more medications to achieve control (<200 mg/dL)
* At lease one of the following metabolic criteria:

  * Fasting blood glucose level > 100 mg/dL
  * Glucose level > 140 mg/dL
  * Diagnosis of type 2 diabetes
* Waist circumference ≥ 102 cm for men or ≥88 cm for women

Exclusion Criteria:

* Stroke/MI/unstable cardiovascular disease within 6 months
* Clinically significant renal, hepatic or psychiatric disease
* Unstable thyroid disease or replacement therapy
* Nephrolithiasis
* Obesity of known genetic or endocrine origin
* Participation in a formal weight loss program or lifestyle intervention
* Glaucoma or intraocular pressure
* Pregnancy or breastfeeding
* Drug or Alcohol abuse
* Smoking cessation within previous 3 months or plans to quit smoking during study
* Eating disorders
* Cholelithiasis within past 6 months
* Excluded medications
* Type 1 diabetes or use of any antidiabetic medication other than metformin
* Previous bariatric surgery
* Bipolar disorder or psychosis
* Steroid hormone therapy
* Systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg
* Creatinine clearance < 60 mL/minute

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2487 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Peterson, Study Director — VIVUS LLC; Kishore Gadde, MD, Study Chair — Duke University
Locations (6):
- United States (6):
  - Research Site, Birmingham, Alabama
  - Research Site, Ridgefield, Connecticut
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Toledo, Ohio
  - Research Site, Austin, Texas

REFERENCES:
- [Derived] Guo F, Garvey WT. Cardiometabolic Disease Staging Predicts Effectiveness of Weight-Loss Therapy to Prevent Type 2 Diabetes: Pooled Results From Phase III Clinical Trials Assessing Phentermine/Topiramate Extended Release. Diabetes Care. 2017 Jul;40(7):856-862. doi: 10.2337/dc17-0088. Epub 2017 Apr 28. PMID 28455281
- [Derived] Garvey WT, Ryan DH, Bohannon NJ, Kushner RF, Rueger M, Dvorak RV, Troupin B. Weight-loss therapy in type 2 diabetes: effects of phentermine and topiramate extended release. Diabetes Care. 2014 Dec;37(12):3309-16. doi: 10.2337/dc14-0930. Epub 2014 Sep 23. PMID 25249652
- [Derived] Gadde KM, Allison DB, Ryan DH, Peterson CA, Troupin B, Schwiers ML, Day WW. Effects of low-dose, controlled-release, phentermine plus topiramate combination on weight and associated comorbidities in overweight and obese adults (CONQUER): a randomised, placebo-controlled, phase 3 trial. Lancet. 2011 Apr 16;377(9774):1341-52. doi: 10.1016/S0140-6736(11)60205-5. Epub 2011 Apr 8. PMID 21481449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at investigative sites in the US between November 2007 through May 2008
Groups:
- VI-0521 Mid: 7.5 mg/46 mg phentermine/topiramate
- VI-0521 Top: 15 mg/92 mg phentermine/topiramate
Period: Overall Study
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top
Started | 994 | 498 | 995
Completed | 616 | 374 | 733
Not Completed | 378 | 124 | 262
Not completed — Adverse Event | 34 | 21 | 67
Not completed — Lost to Follow-up | 132 | 44 | 78
Not completed — Withdrawal by Subject | 151 | 40 | 83
Not completed — Lack of Efficacy | 31 | 1 | 3
Not completed — Pregnancy | 0 | 1 | 2
Not completed — non compliance | 4 | 0 | 11
Not completed — Requirement for restricted medication | 8 | 7 | 5
Not completed — Other | 18 | 10 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top | Total
Number analyzed (Participants) | 994 | 498 | 995 | 2487
Age Continuous [Mean (Standard Deviation); unit: years] | 51.2 (10.3) | 51.1 (10.4) | 51 (10.7) | 51.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 695 | 349 | 693 | 1737
  Male | 299 | 149 | 302 | 750
Region of Enrollment [Number; unit: participants]
  United States | 994 | 498 | 995 | 2487

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Loss From Baseline to Week 56
Time Frame: Baseline to 56 weeks
Population: intent-to-treat last-observation-carried-forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: percent weight loss
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top
Number analyzed (Participants) | 979 | 488 | 981
percent weight loss | 1.24 (0.277) | 7.81 (0.365) | 9.84 (0.275)
Statistical Analysis 1: Comparison: Placebo vs VI-0521 Top; With at least 500 subjects in each of the 3 arms in this trial, the trial has more than 90% power to detect a difference of at least 3.1% between combination and placebo treatment assuming a standard deviation of 5.3% and a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [7.96 to 9.25], Standard Error of Mean 0.328
Statistical Analysis 2: Comparison: Placebo vs VI-0521 Mid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 6.58, 95% CI 2-sided [5.79 to 7.37], Standard Error of Mean 0.403
Statistical Analysis 3: Comparison: VI-0521 Mid vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Intersection-union method applied in a step-down testing approach; Mean Difference (Final Values) = 2.03, 95% CI 2-sided [1.24 to 2.82], Standard Error of Mean 0.402

2. Primary Outcome: Percentage of Subjects With a Weight Loss of at Least 5% at Week 56 With LOCF
Time Frame: Baseline to 56 weeks
Population: intent-to-treat last-observation-carried-forward (ITT-LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top
Number analyzed (Participants) | 979 | 488 | 981
percentage of participants | 20.8 | 62.1 | 70
Statistical Analysis 1: Comparison: Placebo vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 9.03, 95% CI 2-sided [7.34 to 11.11], Standard Error of Mean 0.955
Statistical Analysis 2: Comparison: Placebo vs VI-0521 Mid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 6.27, 95% CI 2-sided [4.93 to 7.97], Standard Error of Mean 0.768
Statistical Analysis 3: Comparison: VI-0521 Mid vs VI-0521 Top; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0018, Regression, Logistic — Intersection-union method applied in a step-down testing approach; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.15 to 1.81], Standard Error of Mean 0.169

ADVERSE EVENTS:
Time Frame: AEs were collected from when written informed consent was provided through 28 days after the last dose of investigational product.
Description: Only subjects who received at least one dose of study drug were included in the safety analysis.
Arm/Group | Placebo | VI-0521 Mid | VI-0521 Top
Serious Adverse Events (participants affected / at risk) | 40/993 | 15/498 | 50/994
Other Adverse Events (participants affected / at risk) | 761/993 | 424/498 | 874/994
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=993) | VI-0521 Mid (N=498) | VI-0521 Top (N=994)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
anemia post-operative (Injury, poisoning and procedural complications) | 1 | 0 | 0
coronary artery disease (Cardiac disorders) | 4 | 0 | 1
myocardial ischemia (Cardiac disorders) | 1 | 0 | 0
urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
transient ischemic attack (Nervous system disorders) | 1 | 0 | 0
brain stem infarction (Nervous system disorders) | 1 | 0 | 0
cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
syncope (Nervous system disorders) | 2 | 0 | 1
hypertension (Vascular disorders) | 1 | 0 | 1
cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
catheter related complications (General disorders) | 1 | 0 | 0
colitis (Gastrointestinal disorders) | 1 | 0 | 0
non-cardiac chest pain (General disorders) | 2 | 0 | 1
chest pain (General disorders) | 2 | 0 | 2
colitis ischemic (Gastrointestinal disorders) | 1 | 0 | 0
diverticulitis (Infections and infestations) | 1 | 2 | 0
small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
invtervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
gastroenteritis (Infections and infestations) | 1 | 0 | 0
arthraligia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
headache (Nervous system disorders) | 1 | 0 | 0
myocardial infarction (Cardiac disorders) | 0 | 1 | 2
hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
hypotension (Vascular disorders) | 0 | 1 | 1
dizziness (Nervous system disorders) | 0 | 1 | 0
tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
brain mass (Nervous system disorders) | 0 | 1 | 0
tachycardia (Cardiac disorders) | 0 | 1 | 0
bursitis infective (Infections and infestations) | 0 | 1 | 0
goiter (Endocrine disorders) | 0 | 1 | 0
umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
esophageal spasm (Gastrointestinal disorders) | 0 | 0 | 1
appendicitis (Infections and infestations) | 0 | 0 | 3
cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
cellulitis (Infections and infestations) | 0 | 0 | 3
skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2
clostridial infection (Infections and infestations) | 0 | 0 | 1
lobar pneumonia (Infections and infestations) | 0 | 0 | 1
drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
gastric ulcer hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
pneumonia (Infections and infestations) | 0 | 0 | 1
incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1
cerebral infarction (Nervous system disorders) | 0 | 0 | 1
intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
liver function test abnormal (Investigations) | 0 | 0 | 1
vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2
fatigue (General disorders) | 0 | 0 | 1
bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
angina pectoris (Cardiac disorders) | 0 | 0 | 1
coital bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=993) | VI-0521 Mid (N=498) | VI-0521 Top (N=994)
Upper Respiratory Tract Infection (Infections and infestations) | 128 | 61 | 133
Nasopharyngitis (Infections and infestations) | 86 | 53 | 98
sinusitis (Infections and infestations) | 67 | 34 | 85
bronchitis (Infections and infestations) | 43 | 22 | 52
urinary tract infection (Infections and infestations) | 37 | 26 | 54
constipation (Gastrointestinal disorders) | 59 | 75 | 173
dry mouth (Gastrointestinal disorders) | 24 | 67 | 207
nausea (Gastrointestinal disorders) | 42 | 18 | 68
diarrhea (Gastrointestinal disorders) | 48 | 32 | 58
headache (Nervous system disorders) | 90 | 35 | 101
paresthesia (Nervous system disorders) | 20 | 68 | 204
dizziness (Nervous system disorders) | 31 | 36 | 99
dysgeusia (Nervous system disorders) | 11 | 37 | 103
back pain (Musculoskeletal and connective tissue disorders) | 49 | 28 | 72
arthralgia (Musculoskeletal and connective tissue disorders) | 54 | 23 | 44
insomnia (Psychiatric disorders) | 47 | 29 | 102
fatigue (General disorders) | 50 | 22 | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.